CLINICAL TRIAL: NCT05294432
Title: Preliminary Validation of the Integral of Pain Relief as a Measure of Pain Relief in Chronic Pain Patients
Brief Title: Validation of the Pain Relief Measure
Status: Completed | Type: Observational
Sponsor: Wilderman Medical Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 8054-02-2019
Record Dates: First submitted 2022-02-11; First posted 2022-03-24 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
Keywords: Pain Relief; Pain Relief Measurement Tool; Integral of Pain Relief; Chronic Pain Clinical Practice
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group: Patients of Wilderman Medical Clinic diagnosed with symptomatic Osteoarthritis of the Knee who were prescribed with at least one intra-articular corticosteroid injection.

SUMMARY:
The purpose of this study is to provide evidence for the empirical and clinical utility of a novel pain relief measure, the IPR, dimensions of which will be validated against the present gold standards for pain measurement.

DETAILED DESCRIPTION:
There are a number of validated unidimensional and multidimensional tools used to measure pain levels. The present widely used in clinical practice standard measure of pain relief in patients experiencing acute or chronic pain is a change in the numerical rating scale (NRS) score. NRS is a unidimensional scale that requires patients to mark their pain level from 0 (no pain) to 10 (worst pain). The NRS provides practitioners with pain levels pre-and-post treatment and is used as an indication of treatment efficacy. A significant limitation of the NRS, however, is that it provides an estimation of a single dimension of pain, pain intensity. Pain and pain relief, on the other hand, may have many dimensions including pain intensity, duration and magnitude of pain relief. Current multidimensional measures fail to capture duration of pain relief, thus there is a necessity to improve pain assessment tools. The integral of pain relief (IPR) is a novel two-dimensional measure of pain relief and duration of pain relief following treatment and may provide a more accurate depiction of post-treatment pain as well as intervention effectiveness. In this prospective cohort study, we intend to assess the validity of the IPR using validated measures of change in pain intensity (NRS), and the Patients' Global Impression of Change (PGIC) as well as The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) in patients treated with corticosteroid injections for the osteoarthritis of knee joint.

The primary objectives of this study include:

* Compare pre- and post-treatment scores of the i) IPR dimensions (post-treatment), ii) NRS (pre- and post-treatment), iii) PGIC (post-treatment), and iv) WOMAC (pre- and post-treatment) in patients with knee osteoarthritis treated with intra-articular corticosteroid injections.
* Provide preliminary validation for the Integral of Pain Relief as a clinical assessment tool of post-treatment pain relief and treatment efficacy.

Secondary objectives of this study include:

* Assess whether baseline patient characteristics such as pre-treatment pain intensity score, disease-associated pain duration, age, gender, co-morbidity with diabetes, symptoms of either depression or anxiety, or both, litigation status, occupation, and level of education are important predictors to responses on the four pain outcome measures.
* Assess patients' impression of their usage of the daily pain diary versus providing the percentage and duration of pain relief at follow up time points.

ELIGIBILITY:
Inclusion Criteria:

* Given written Informed Consent to participate in the study
* Male or female ≥40 years of age
* Diagnosis of unilateral or bilateral OA of the knee for at least 6 months prior to Screening requiring the use of regular therapies.
* If bilateral OA exists, pain in the contralateral knee must be less than pain in the index knee as reported by patient
* Index knee pain on most days (>15) over the last month
* Mean score of ≥4 and ≤9 on the 24-hr average pain score (0-10 NRS) using the average daily ratings at least 5 out of 7 days prior to Day 1(Baseline)
* Have been prescribed and scheduled to receive at least one corticosteroid (triamcinolone) injection to the affected knee
* Willingness and ability to comply with the study procedures and visit schedules and the ability to follow verbal and written instructions

Exclusion Criteria:

* Lack of signed Informed Consent Form
* Age less than 40 years old
* Have any contraindications to administration of corticosteroid medication by intra-articular injection
* Patients with diagnoses of fibromyalgia, chronic pain syndrome, or other concurrent medical or arthritic conditions which could interfere with the evaluation of the index knee
* Patients with diagnoses of rheumatoid arthritis, psoriatic arthritis, or any other form of inflammatory arthritis
* Planned/anticipated surgery in the affected area within 3 months during the study period.
* Previous intra-articular corticosteroid injection into the index joint within 3 months prior to Screening
* Concomitant treatment with corticosteroid or other injections into the index joint (e.g. prolotherapy) within 3 months during the study period
* Concomitant treatment with oral or topical (to the index knee) corticosteroids within 3 months during the study period (except inhaled, intranasal, or topical applied not to the index knee)
* Any other investigational drug/biologic applied to affected area within 3 months during the study period
* Diagnosis of dementia or other cognitive impairments that would preclude questionnaires completion
* Any clinically significant acute or chronic medical conditions that, in the judgment of Investigator, would preclude the use of corticosteroid injections or that could compromise patient safety, limit the patient's ability to complete the study, and/or compromise the objectives of the study
* Participation in any other clinical study within 3 months prior to Screening and during the study period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Wilderman Medical Clinic ≥40 years of age diagnosed with symptomatic Osteoarthritis of the Knee who are prescribed at least one corticosteroid intra-articular injection into the knee.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Integral of Pain Relief (dimensions) | Post-interventional at week 2
  Patient's reported percentage (%) and duration of pain relief (days)
Integral of Pain Relief (dimensions) | Post-interventional at week 4
  Patient's reported percentage (%) and duration of pain relief (days)
Integral of Pain Relief (dimensions) | Post-interventional at week 6
  Patient's reported percentage (%) and duration of pain relief (days)
Integral of Pain Relief (dimensions) | Post-interventional at week 8
  Patient's reported percentage (%) and duration of pain relief (days)
Integral of Pain Relief (dimensions) | Post-interventional at week 12
  Patient's reported percentage (%) and duration of pain relief (days)
Change in Pain Intensity Numeric Rating Scale (NRS) score | Baseline, post-interventional at week 2
  Change in average daily (24-hr) pain intensity scores (NRS) from baseline to 2 weeks post-interventional. Numeric Rating Scale pain intensity score is recorded daily via pain diary starting from day -7 (one week before baseline). Numeric Rating Scale pain intensity score is recorded daily via pain diary. Numeric Rating Scale is a one-dimensional measure of pain intensity. The pain intensity is rated by participant using a scale from 0 to 10, 0 being the least (no pain) to 10 (worst pain imaginable).
Pain Intensity Numeric Rating Scale | Baseline, post-interventional at week 4
  Change in average daily (24-hr) pain intensity scores from baseline to 4 weeks post-interventional. Numeric Rating Scale pain intensity score is recorded daily via pain diary starting from day -7 (one week before baseline). Numeric Rating Scale pain intensity score is recorded daily via pain diary. Numeric Rating Scale is a one-dimensional measure of pain intensity. The pain intensity is rated by participant using a scale from 0 to 10, 0 being the least (no pain) to 10 (worst pain imaginable).
Pain Intensity Numeric Rating Scale (NRS) | Baseline, post-interventional at week 6
  Change in average daily (24-hr) pain intensity scores (NRS) from baseline to 6 weeks post-interventional. Numeric Rating Scale pain intensity score is recorded daily via pain diary starting from day -7 (one week before baseline). Numeric Rating Scale pain intensity score is recorded daily via pain diary. Numeric Rating Scale is a one-dimensional measure of pain intensity. The pain intensity is rated by participant using a scale from 0 to 10, 0 being the least (no pain) to 10 (worst pain imaginable).
Pain Intensity Numeric Rating Scale (NRS) | Baseline, post-interventional at week 8
  Change in average daily (24-hr) pain intensity scores (NRS) from baseline to 8 weeks post-interventional. Numeric Rating Scale pain intensity score is recorded daily via pain diary starting from day -7 (one week before baseline). Numeric Rating Scale pain intensity score is recorded daily via pain diary. Numeric Rating Scale is a one-dimensional measure of pain intensity. The pain intensity is rated by participant using a scale from 0 to 10, 0 being the least (no pain) to 10 (worst pain imaginable).
Pain Intensity Numeric Rating Scale (NRS) | Baseline, post-interventional at week 12
  Change in average daily (24-hr) pain intensity scores (NRS) from baseline to 12 weeks post-interventional. Numeric Rating Scale pain intensity score is recorded daily via pain diary starting from day -7 (one week before baseline). Numeric Rating Scale pain intensity score is recorded daily via pain diary. Numeric Rating Scale is a one-dimensional measure of pain intensity. The pain intensity is rated by participant using a scale from 0 to 10, 0 being the least (no pain) to 10 (worst pain imaginable).
Western Ontario and McMaster Universities (WOMAC® 3.1) Osteoarthritis Index | Baseline, post-interventional at weeks 2
  Change in total score from baseline to 2 weeks post-interventional. Western Ontario and McMaster Universities (WOMAC® 3.1) Osteoarthritis Index is a Likert 5 point scale for pain, stiffness and function domains. Activities in each domain are rated by a study participant according to the following scale of difficulty: 0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely.
Western Ontario and McMaster Universities (WOMAC® 3.1) Osteoarthritis Index | Baseline, post-interventional at week 4
  Change in total score from baseline to 4 weeks post-interventional. Western Ontario and McMaster Universities (WOMAC® 3.1) Osteoarthritis Index is a Likert 5 point scale for pain, stiffness and function domains. Activities in each domain are rated by a study participant according to the following scale of difficulty: 0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely.
Western Ontario and McMaster Universities (WOMAC® 3.1) Osteoarthritis Index | Baseline, post-interventional at week 6
  Change in total score from baseline to 6 weeks post-interventional. Western Ontario and McMaster Universities (WOMAC® 3.1) Osteoarthritis Index is a Likert 5 point scale for pain, stiffness and function domains. Activities in each domain are rated by a study participant according to the following scale of difficulty: 0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely.
Western Ontario and McMaster Universities (WOMAC® 3.1) Osteoarthritis Index | Baseline, post-interventional at week 8
  Change in total score from baseline to 8 weeks post-interventional. Western Ontario and McMaster Universities (WOMAC® 3.1) Osteoarthritis Index is a Likert 5 point scale for pain, stiffness and function domains. Activities in each domain are rated by a study participant according to the following scale of difficulty: 0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely.
Western Ontario and McMaster Universities (WOMAC® 3.1) Osteoarthritis Index | Baseline, post-interventional at week 12
  Change in total score from baseline to 12 weeks post-interventional. Western Ontario and McMaster Universities (WOMAC® 3.1) Osteoarthritis Index is a Likert 5 point scale for pain, stiffness and function domains. Activities in each domain are rated by a study participant according to the following scale of difficulty: 0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely.
Patient's Global Impression of Change (PGIC) | Post-interventional at week 2
  Patient's Global Impression of Change (PGIC) scores from Baseline to 2 weeks post-interventional. Patient's Global Impression of Change (PGIC) is a 7-point single item scale ranging from "very much worse" to "very much improved" with "no change" with "no change" at mid-point that evaluated improvement in overall status with treatment during clinical trial.
Patient's Global Impression of Change (PGIC) | Post-interventional at week 4
  Patient's Global Impression of Change (PGIC) scores from Baseline to 4 weeks post-interventional. Patient's Global Impression of Change (PGIC) is a 7-point single item scale ranging from "very much worse" to "very much improved" with "no change" with "no change" at mid-point that evaluated improvement in overall status with treatment during clinical trial.
Patient's Global Impression of Change (PGIC) | Post-interventional at week 6
  Patient's Global Impression of Change (PGIC) scores from Baseline to 6 weeks post-interventional. Patient's Global Impression of Change (PGIC) is a 7-point single item scale ranging from "very much worse" to "very much improved" with "no change" with "no change" at mid-point that evaluated improvement in overall status with treatment during clinical trial.
Patient's Global Impression of Change (PGIC) | Post-interventional at week 8
  Patient's Global Impression of Change (PGIC) scores from Baseline to 8 weeks post-interventional. Patient's Global Impression of Change (PGIC) is a 7-point single item scale ranging from "very much worse" to "very much improved" with "no change" with "no change" at mid-point that evaluated improvement in overall status with treatment during clinical trial.
Patient's Global Impression of Change (PGIC) | Post-interventional at week 12
  Patient's Global Impression of Change (PGIC) scores from Baseline to 12 weeks post-interventional. Patient's Global Impression of Change (PGIC) is a 7-point single item scale ranging from "very much worse" to "very much improved" with "no change" with "no change" at mid-point that evaluated improvement in overall status with treatment during clinical trial.

SECONDARY OUTCOMES:
Use of Analgesic Medication | Baseline, Post-intervention at week 2
  Change in average consumption of analgesic medication (days) as per patient's daily diary from baseline to 2 weeks post-interventional.
Use of Analgesic Medication | Baseline, Post-intervention at week 4
  Change in average consumption of analgesic medication (days) as per patient's daily diary from baseline to 4 weeks post-interventional.
Use of Analgesic Medication | Baseline, Post-intervention at week 6
  Change in average consumption of analgesic medication (days) as per patient's daily diary from baseline to 6 weeks post-interventional.
Use of Analgesic Medication | Baseline, Post-intervention at week 8
  Change in average consumption of analgesic medication (days) as per patient's daily diary from baseline to 8 weeks post-interventional.
Use of Analgesic Medication | Baseline, Post-intervention at week 12
  Change in average consumption of analgesic medication (days) as per patient's daily diary from baseline to 12 weeks post-interventional.
Patient's Survey | Post-interventional at 12 weeks
  Patient's impression on completing daily pain diary versus providing percentage and duration of pain relief

CONTACTS AND LOCATIONS:
Overall Officials: Igor Wilderman, MD, Principal Investigator — Wilderman Medical Clinic
Locations (1):
- Wilderman Medical Clinic, Thornhill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided